CLINICAL TRIAL: NCT06093971
Title: Remimazolam Versus Propofol for General Anesthesia Induction in Patients on Renin-angiotensin System Blockers Undergoing Robot-assisted Laparoscopic Prostatectomy: A Randomized Controlled Study
Brief Title: Remimazolam Versus Propofol for General Anesthesia Induction in Patients on Renin-angiotensin System Blockers Undergoing Robot-assisted Laparoscopic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2023-0803
Record Dates: First submitted 2023-09-12; First posted 2023-10-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Prostate Tumor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group remimazolam (Experimental): During anesthesia induction, the remimazolam group (group R) receives remimazolam (0.2 mg/kg). If necessary, an additional dose of remimazolam (0.1 mg/kg) is administered.
  Interventions: Drug: remimazolam
- Group propofol (Active Comparator): During anesthesia induction, the propofol group (group P) receives propofol (1.0 mg/kg). If necessary, an additional dose of propofol (0.5 mg/kg) is administered.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: remimazolam — Remimazolam is administered for anesthesia induction.
  Arms: Group remimazolam
Drug: Propofol — Propofol is administered for anesthesia induction.
  Arms: Group propofol

SUMMARY:
The investigators conduct a random assignment into either the remimazolam group or the propofol group. Depending on the group assignment, either remimazolam (0.2 mg/kg) or propofol (1.0 mg/kg) is administered. If necessary, additional doses of remimazolam (0.1 mg/kg) or propofol (0.5 mg/kg) are given. The standard anesthesia procedure of our institution is followed, and blood pressure data recorded during the surgery is analyzed (mean arterial pressure <65mmHg is defined as hypotension).

ELIGIBILITY:
Inclusion Criteria:

Patients who undergo robot-assisted laparoscopic prostatectomy and who have taken renin-angiotensin system blockers for more than 3 months.

Exclusion Criteria:

1. emergency surgery
2. If the subject includes those who cannot read the consent form (e.g. illiterate, foreigners, etc.)
3. cognitive dysfunction
4. Atrial fibrillation, moderate to severe valvular disease, ejection fraction of 35% or less
5. Patients who did not take renin-angiotensin system blockers on the day of surgery

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Hypotension occurrence (unit: number of patients) | during the total anesthesia duration
  "MAP<65mmHg for 1 min
Amount of hypotension (unit: mmHg) | during the total anesthesia duration
  time-weighted average MAP <65mmHg => depth of hypotension (mmHg) below a MAP of 65 mmHg * time (min) below a MAP of 65 mmHg)/ total duration of surgery (min)
Vasopressor dose (unit: mcg for norepinephrine) | during the total anesthesia duration
  total dose of norepinephrine administered
Vasopressor dose (unit for vasopressin) | during the total anesthesia duration
  total dose of vasopressin administered

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HJ, Kim N, Kim J, Park JH, Shin HJ, Yang J, Kim SY. Intraoperative hypotension after remimazolam or propofol induction with sevoflurane maintenance in angiotensin II receptor blockers-treated patients: a randomized controlled trial. Sci Rep. 2025 Nov 13;15(1):39805. doi: 10.1038/s41598-025-23469-y. PMID 41233396